CLINICAL TRIAL: NCT07065812
Title: The Impact of Team Familiarity on Surgical Outcomes and Patient Safety in Non-Cardiac Surgery
Brief Title: Team Familiarity and Perioperative Outcomes in Non-Cardiac Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Peng Zhendan, Attending physician, Zhongda Hospital
Other Study IDs: 2025ZDSYLL172-P01
Record Dates: First submitted 2025-06-06; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Operating Room Efficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surgical team familiarity — Surgical team familiarity: the degree of collaboration within the surgical team is statistically described based on data regarding team personnel and composition, which is used to calculate the Intraoperative Familiarity Score (IFS)-the core component of this study. The specific methodology includes IFS=（X1+X2+X3+X4+X5+X6…）/ N N=nCr=n!/r!(n-r)! Here, X represents the number of times a pair of team members has worked together over a specified period (this process is repeated for all possible pairings in the team), and N is the total number of possible pairwise combinations in the team.
Other: Composition and Dynamics of the Surgical Team — Basic indicators reflecting surgical team personnel and composition:
  1. Number of surgical, anesthesia, and nursing team members participating in procedures: are obtainable via the Anesthesia Information Management System (AIMS).
  2. Shift changes among surgical, anesthesia, and nursing teams during individual procedures: can be tracked through the AIMS.
  3. Gender ratio within surgical, anesthesia, and nursing teams: will be derived from the Hospital Information System (HIS)."

SUMMARY:
The goal of this retrospective observational study is to quantify the impact of team collaboration on work efficiency in operating room and patient safety outcomes in non-cardiac surgical teams. The main purpose is to answer:

How does team collaboration affect work efficiency in operating room and patient safety outcomes during/after surgery? The data will be obtained from the Hospital Electronic Medical Record Information System, participants already finished all the planned surgeries.

DETAILED DESCRIPTION:
This study aims to reveal the crucial role of teamwork in surgical operations. Firstly, by calculating the degree of collaboration within the surgical team, we quantify the interactions, communication, and trust among team members, and subsequently analyze the impact of this collaboration on surgical team work efficiency indicators including pre-anesthesia preparation time, anesthesia induction time, and operation time, to identify optimal practices. Secondly, it analyzes how the degree of cooperation among surgical teams affects patient safety indicators such as intraoperative blood loss, the incidence of unplanned secondary surgeries, and the in-hospital mortality rate, thereby revealing the direct or indirect contribution of teamwork to patient safety. The impact of surgical team size, gender composition, and shift patterns on work efficiency and patient safety indicators was also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* All elective surgeries for adults (age ≥18 years)

Exclusion Criteria:

* Surgeries in which patient demographics (age, gender), ASA grade, procedure details, and positional data were unattainable
* Cardiac surgical procedures (with a fixed surgical team)
* Operations under non-intubated general anesthesia or intravenous anesthesia (primarily diagnostic procedures not requiring close multidisciplinary collaboration)
* Surgical cases with missing data on pre-anesthesia preparation time, anesthesia induction time, and surgical procedure duration
* Surgical cases with missing data on team members' years of experience and gender information.
* Surgical cases with missing data on intra- and post-operative major complications and other safety-related outcome measures

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes elective surgical patients who underwent procedures at Zhongda Hospital Southeast University between January 1, 2016, and March 31, 2025, and their respective surgical team members.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Surgical Team Efficiency | Perioperative
  The primary outcome measure of this study is surgical team efficiency, which is represented by three time intervals: pre-anesthesia preparation time (from patient entry into the operating room to anesthesia initiation), anesthesia induction time (from anesthesia initiation to surgery start), and surgical duration (from surgery start to surgery end). These intervals are calculated in minutes using the anesthesia information management system (AIMS), with timestamps recorded in the anesthesia record form within AIMS for the following key events: patient arrival in the operating room, anesthesia initiation, surgery start, surgery conclusion, anesthesia end and patient exit from the operating room.

SECONDARY OUTCOMES:
Blood loss | Perioperative
  The total volume of blood loss during the procedure，measured in milliliters (mL) .
Duration of PACU (Post-Anesthesia Care Unit) stay | Perioperative
  From admission to discharge from the PACU recorded in minutes/hours
Unplanned ICU admission within 24 hours post-surgery | Perioperative
Number of postoperative ICU admissions | Perioperative
ICU stay duration recorded in days | Perioperative
Unplanned secondary surgery | Perioperative
Postoperative infection | Perioperative
In-hospital mortality | Perioperative
Total hospital stay duration recorded in days | Perioperative
Total hospitalization expenses recorded in RMB/CNY | Perioperative
Improvement status of the primary diagnosis on the day of discharge | Perioperative
Rescue events during hospitalization | Perioperative